CLINICAL TRIAL: NCT06336460
Title: Pericapsular Nerve Group (PENG) Block vs. the Fascia Iliaca Compartment (FIC) Block for Patients With Isolated Hip Fractures in the Emergency Department
Brief Title: PENG vs. FIC Blocks in Hip Fractures in the ED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orange Park Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-537
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Hip Fractures; Nerve Block; Analgesia
MeSH Terms: conditions — Hip Fractures; Agnosia | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The research associate/outcome assessor will not have access to group assignment and will therefore be blinded to the type of block. Although the patient, their caregiver(s), and the clinician caring for the patient will not be directly informed of the group assignment, a note will be logged in the clinical record by the physician placing the block indicating the details of the block after this procedure has been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pericapsular Nerve Group (PENG) Block (Experimental)
  Interventions: Procedure: Pericapsular Nerve Group (PENG) Block
- Fascia Iliaca Compartment (FIC) Block (Experimental)
  Interventions: Procedure: Fascia Iliaca Compartment (FIC) Block for Patients with Isolated Hip Fractures

INTERVENTIONS:
Procedure: Pericapsular Nerve Group (PENG) Block — Under sterile technique, physician will identify relevant landmarks including the femoral artery, femoral vein, femoral nerve, ileopubic eminence (IPE), anterior inferior iliac spine (AIIS), psoas tendon (PT). Target area is bony space between AIIS and IPE adjacent to PT.
  Using in-plane technique with constant visualization, needle will be inserted through skin and soft tissue targeting fascial plane below the psoas tendon, above ilium bone. Landmark lies between the AIIS and IPE, just lateral to psoas tendon.
  As needle tip reaches target, small volume of normal saline will be injected to hydrodissect tissue. Fluid will start to spread along fascial plane, lifting the psoas tendon from ilium, confirming proper positioning.
  Normal saline will then be switched to anesthetic (30mL of Bupivacaine 0.25%).
  After full volume of anesthetic has been injected, a small volume (5mL) of normal saline will be injected to flush line of remaining anesthetic. Needle will then be withdrawn.
  Arms: Pericapsular Nerve Group (PENG) Block
Procedure: Fascia Iliaca Compartment (FIC) Block for Patients with Isolated Hip Fractures — Under sterile technique, physician will identify relevant landmarks, including femoral artery, femoral vein, femoral nerve, iliacus muscle with overlying fascia iliaca.
  Using in-plane technique with constant visualization, needle will be inserted through skin and soft tissue targeting the fascial plane above iliacus muscle.
  As needle tip reaches the target, a small volume of normal saline will be injected to hydrodissect tissue. Fluid will start to spread along fascial plane, confirming proper positioning.
  Normal saline will then be switched to anesthetic (30mL of Bupivacaine 0.25%).
  After full volume of anesthetic has been injected, a small volume (5mL) of normal saline will be injected to flush the line of remaining anesthetic. The needle will then be withdrawn.
  Arms: Fascia Iliaca Compartment (FIC) Block

SUMMARY:
This study is a prospective, randomized clinical trial assessing the efficacy of physician-performed ultrasound-guided pericapsular nerve group (PENG) block vs fascia iliaca compartment (FIC) block for pain control in acute hip fracture.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>= 18 years of age)
* Isolated proximal hip fracture (defined as Intertrochanteric or more proximal) as identified by X-ray, Computed Tomography (CT) scan or Magnetic Resonance Imaging (MRI) scan
* Glasgow Coma Score (GCS) = 15
* Subjective pain score of >= 5 on a scale of 0 to 10 just prior to the nerve block placement

Exclusion Criteria:

* Patients who are unable to give consent due to altered mental status or dementia
* Clinically intoxicated patients
* Patients who are unable to communicate their numeric level of pain
* Open fracture or penetrating hip trauma
* Signs of infection or laceration at injection site
* Patients with multi-system trauma
* Painful distracting injury (injury causing significant pain that distracts the patient from having reliable scoring of hip fracture pain, e.g. humerus fracture, dislocated joint)
* Requiring immediate surgical intervention (< 1 hour)
* Deemed clinically unstable by treating physician
* Abnormal vital signs (Pulse>120bpm, Systolic blood pressure < 100 mm Hg, Pulse O2 < 95%)
* Patients on long-acting systemic opioid analgesia
* Allergy to amide local anesthetics
* Vulnerable populations including pregnant patients, prisoners, children, elderly dementia patients. All precautions will be taken to avoid coercion, harm and exploitation of these vulnerable populations, thus they are to be excluded from this study. They will receive pain medications as deemed appropriate by their treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Numeric pain score at 30 minutes | 30 minutes after block placement
Numeric pain score at 60 minutes | 1 hour after block placement

SECONDARY OUTCOMES:
Cumulative Morphine Milligram Equivalents in 24 hours after enrollment | 24 hours after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Taryn Hoffman, MD, Principal Investigator — HCA Florida Orange Park Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhoi S, Chandra A, Galwankar S. Ultrasound-guided nerve blocks in the emergency department. J Emerg Trauma Shock. 2010 Jan;3(1):82-8. doi: 10.4103/0974-2700.58655. PMID 20165729
- [Background] Pasquier M, Taffe P, Hugli O, Borens O, Kirkham KR, Albrecht E. Fascia iliaca block in the emergency department for hip fracture: a randomized, controlled, double-blind trial. BMC Geriatr. 2019 Jul 1;19(1):180. doi: 10.1186/s12877-019-1193-0. PMID 31262265
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Luftig J, Dreyfuss A, Mantuani D, Howell K, White A, Nagdev A. A new frontier in pelvic fracture pain control in the ED: Successful use of the pericapsular nerve group (PENG) block. Am J Emerg Med. 2020 Dec;38(12):2761.e5-2761.e9. doi: 10.1016/j.ajem.2020.05.085. Epub 2020 May 28. PMID 32532621
- [Background] Marrone F, Graziano G, Paventi S, Tomei M, Gucciardino P, Bosco M. Analgesic efficacy of Pericapsular Nerve Group (PENG) block compared with Fascia Iliaca Block (FIB) in the elderly patient with fracture of the proximal femur in the emergency room. A randomised controlled trial. Rev Esp Anestesiol Reanim (Engl Ed). 2023 Nov;70(9):501-508. doi: 10.1016/j.redare.2022.10.010. Epub 2023 Sep 6. PMID 37678449
- [Background] Aliste J, Layera S, Bravo D, Jara A, Munoz G, Barrientos C, Wulf R, Branez J, Finlayson RJ, Tran Q. Randomized comparison between pericapsular nerve group (PENG) block and suprainguinal fascia iliaca block for total hip arthroplasty. Reg Anesth Pain Med. 2021 Oct;46(10):874-878. doi: 10.1136/rapm-2021-102997. Epub 2021 Jul 20. PMID 34290085